CLINICAL TRIAL: NCT01696526
Title: Bioefficiency of of Conventional Fish and Vitamin D Fortified Fish in Healthy Volunteers
Brief Title: Bioefficiency of of Conventional Fish and Vitamin D Fortified Fish
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ulrike Lehmann (Other)
Responsible Party: Sponsor-Investigator, Ulrike Lehmann, Scientist, Martin-Luther-Universität Halle-Wittenberg
Organization: Martin-Luther-Universität Halle-Wittenberg (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: BMBF 0315668
Record Dates: First submitted 2012-09-27; First posted 2012-10-01 (Estimated); Last update posted 2012-12-20 (Estimated); Status verified 2012-12

CONDITIONS: Vitamin D Deficiency
Keywords: vitamin D; bioeffiency; vitamin d fortified fish
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Methods

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- vitamin D fortified fish (Experimental): Human volunteers receiving vitamin D fortified fish, 4 weeks
  Interventions: Other: vitamin D fortified fish
- conventional fish (Placebo Comparator): consumption of conventional fish , 4 weeks
  Interventions: Other: conventional fish

INTERVENTIONS:
Other: vitamin D fortified fish — fish containing vitamin D3
  Other Names: intervention
  Arms: vitamin D fortified fish
Other: conventional fish — fish containing low concentrations of vitamin D3
  Other Names: placebo
  Arms: conventional fish

SUMMARY:
The aim of this study is to investigate the bioavailability of conventional and vitamin D fortified fish as measured by the increase of the specific hydroxy form by 25(OH)D3.

DETAILED DESCRIPTION:
Study design: Human volunteers will receive conventional fish or vitamin D fortified fish for a period of 4 weeks. At baseline and after 4 weeks, 25(OH)D3 will be measured in serum as the main outcome variables. Additional outcome variables are the Ca concentration in serum, PTH concentration in serum.

Groups/Cohorts Assigned Interventions

1. Placebo group receiving conventional fish
2. intervention group receiving vitamin D fortified fish

ELIGIBILITY:
Inclusion Criteria:

* 18 years
* healthy

Exclusion Criteria:

* supplementation of vitamin d and calcium
* hypercalcemia
* hypercalciuria
* chronical illness (diabetes, kidney diseases, cardiovascular diseases)
* serum-creatinine above 115 mmol/l
* pregnancy or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2012-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
change of 25-hydroxvitamin D | after 4 weeks of consumption

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele I. Stangl, Prof., Study Director — Institut für Agrar- und Ernährungswissenschaften
Locations (1):
- Naturwissenschaftliche Fakultät, Halle, Saxony-Anhalt, Germany